CLINICAL TRIAL: NCT00073216
Title: A Phase I Clinical Trial to Evaluate the Safety and Immunogenicity of a Clade B Gag DNA/PLG and Env DNA/PLG Microparticles Vaccine and a Clade B Recombinant, Oligomeric gp140/MF59 Adjuvant Vaccine in Healthy, HIV-1 Uninfected Adult Participants
Brief Title: Safety of and Immune Response to a Combination HIV Vaccine Regimen in HIV Uninfected Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Purpose: Prevention
Other Study IDs: HVTN 049; 10054 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 2003-11-18; First posted 2003-11-19 (Estimated); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: HIV Seronegativity; HIV Preventive Vaccine
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Biological: Clade B gag DNA/PLG and env DNA/PLG Microparticles
Biological: Clade B Recombinant, Oligomeric gp140/MF59 Adjuvant

SUMMARY:
To prevent HIV infection, a vaccine that produces strong HIV-specific humoral (B-cell) and cellular (T-cell) immune system responses is desirable. The purpose of this study is to test the safety of and immune response to a novel combination HIV vaccine in HIV uninfected adults. This study will also test the safety of and immune response to a protein vaccine given alone.

DETAILED DESCRIPTION:
The development of a vaccine eliciting HIV-specific humoral and cellular immune responses is desirable for the prevention of HIV infection. This study will investigate a combination vaccine regimen consisting of priming with DNA followed by boosting with a recombinant envelope glycoprotein adjuvanted in MF59.

All participants will be followed for 15 months. Participants enrolled in Groups 1, 2, 3, and 4 will receive either the vaccine or placebo. Study visits will be completed at initial entry; five visits every 14 days for the first 2.5 months; and visits at Months 4, 4.5, 6, 6.5, 9, 9.5, 12, and 15. All participants will undergo physical exams, urine collection, and blood tests to assess safety, HIV infection, and immune responses to injections. Risk reduction/pregnancy prevention counseling will be given at every study visit. Participants will also be asked to complete questionnaires about outside testing and beliefs at certain visits.

There are two parts to this study. In Part A, participants will be sequentially assigned to one of three groups. Each group will receive injections of different amounts of either DNA vaccine or placebo at entry, Month 1, and Month 2. This is followed by identical injections of glycoprotein/adjuvant or placebo at Months 6 and 9. Group 1 will receive 250 mcg each of the gag and env DNA plasmid with microparticle vaccine; Group 2 will receive 500 mcg of each vaccine; Group 3 will receive 1000 mcg of each vaccine. Participants will be enrolled sequentially from low to high dose beginning with Group 1.

In Part B, Group 4 will begin the second part of the study simultaneously after safety review of all participants in Part A. Group 4 participants will receive identical injections of either DNA vaccine or placebo at entry and at Months 1, 2, 6, and 9.

Group 5 will begin enrollment after enrollment is completed for Groups 1, 2, 3, and 4. Group 5 participants will receive identical injections of either glycoprotein/adjuvant or placebo at study entry and at Months 3 and 9. There will be 11 study visits for Group 5 participants; they will occur at screening, study entry, and Months 0.5, 2, 3, 3.5, 6, 9, 9.5, 12, and 15. A physical exam and risk reduction/pregnancy prevention counseling will occur at all visits; participants will be asked at every visit about any adverse events they may have experienced. Blood and urine collection will occur at selected visits. Participants will be also asked to complete questionnaires about outside testing and beliefs at certain visits.

ELIGIBILITY:
Note: As of 07/01/05, Group 5 will begin enrollment after enrollment into Groups 1, 2, 3, and 4 is completed.

Inclusion Criteria

* Understanding of vaccination procedure
* Willing to receive HIV test results and provide informed consent
* Good general health
* HIV negative
* Hepatitis B surface antigen negative
* Anti-hepatitis C virus (HCV) antibody negative, or negative for HCV PCR if the anti-HCV is positive
* Not pregnant and agrees to use acceptable forms of contraception

Exclusion Criteria

* Received HIV vaccines or placebo in a prior HIV vaccine trial
* Immunosuppressive medications within 168 days prior to study
* Blood products within 120 days prior to study
* Immunoglobulin within 60 days prior to study
* Live attenuated vaccines within 30 days prior to study
* Investigational research agents within 30 days prior to study
* Medically indicated subunit or killed vaccines within 14 days prior to study
* Current anti-tuberculosis prophylaxis or therapy
* Anaphylaxis or other serious adverse reactions to vaccines; a person who had an adverse reaction to pertussis vaccine as a child is not excluded
* Autoimmune disease or immunodeficiency
* Active syphilis infection
* Unstable asthma (e.g., use of oral, orally inhaled, or intravenous corticosteroids, emergent care, urgent care, hospitalization or intubation during the past 2 years)
* Diabetes mellitus; a participant with past gestational diabetes is not excluded
* Thyroid disease, including removal of thyroid and diagnoses requiring medication
* Serious angioedema
* Uncontrolled hypertension
* Diagnosis of bleeding disorder
* Malignancy, except those with a surgical excision and subsequent observation period that in the investigator's estimate has a reasonable assurance of sustained cure and/or is unlikely to recur during the period of the study
* Seizure disorder requiring medication within the last 3 years
* Absence of the spleen
* Mental illness that would interfere with compliance with the protocol
* Breastfeeding
* Unprotected rectal or vaginal sex with a partner known to be HIV infected within 6 months of enrollment

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Safety (local and systemic reactogenicity signs and symptoms, laboratory measures, and adverse and serious experiences)
immunogenicity (presence of HIV-specific immune response as measured by the interferon-gamma ELISpot, FACS Intracellular Cytokine Staining [ICS], neutralizing antibody, or HIV antigen-binding ELISA assays)
social impacts (negative experiences or problems reported by the participants)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Spearman, Study Chair — Vanderbilt University; Michelle Lally, Study Chair — Brown University
Locations (4):
- United States (4):
  - Saint Louis Univ. School of Medicine, HVTU, St Louis, Missouri
  - Miriam Hospital's HVTU, Providence, Rhode Island
  - Vanderbilt Vaccine CRS, Nashville, Tennessee
  - FHCRC/UW Vaccine CRS, Seattle, Washington

REFERENCES:
- [Background] Malkevitch NV, Robert-Guroff M. A call for replicating vector prime-protein boost strategies in HIV vaccine design. Expert Rev Vaccines. 2004 Aug;3(4 Suppl):S105-17. doi: 10.1586/14760584.3.4.s105. PMID 15285710
- [Background] O'Hagan D, Singh M, Ugozzoli M, Wild C, Barnett S, Chen M, Schaefer M, Doe B, Otten GR, Ulmer JB. Induction of potent immune responses by cationic microparticles with adsorbed human immunodeficiency virus DNA vaccines. J Virol. 2001 Oct;75(19):9037-43. doi: 10.1128/JVI.75.19.9037-9043.2001. PMID 11533167
- [Background] O'Hagan DT, Ugozzoli M, Barackman J, Singh M, Kazzaz J, Higgins K, Vancott TC, Ott G. Microparticles in MF59, a potent adjuvant combination for a recombinant protein vaccine against HIV-1. Vaccine. 2000 Mar 6;18(17):1793-801. doi: 10.1016/s0264-410x(99)00522-8. PMID 10699327
- [Background] Slobod KS, Bonsignori M, Brown SA, Zhan X, Stambas J, Hurwitz JL. HIV vaccines: brief review and discussion of future directions. Expert Rev Vaccines. 2005 Jun;4(3):305-13. doi: 10.1586/14760584.4.3.305. PMID 16026246
- [Background] Stratov I, DeRose R, Purcell DF, Kent SJ. Vaccines and vaccine strategies against HIV. Curr Drug Targets. 2004 Jan;5(1):71-88. doi: 10.2174/1389450043490686. PMID 14738219
- [Derived] Spearman P, Lally MA, Elizaga M, Montefiori D, Tomaras GD, McElrath MJ, Hural J, De Rosa SC, Sato A, Huang Y, Frey SE, Sato P, Donnelly J, Barnett S, Corey LJ; HIV Vaccine Trials Network of NIAID. A trimeric, V2-deleted HIV-1 envelope glycoprotein vaccine elicits potent neutralizing antibodies but limited breadth of neutralization in human volunteers. J Infect Dis. 2011 Apr 15;203(8):1165-73. doi: 10.1093/infdis/jiq175. PMID 21451004